CLINICAL TRIAL: NCT01392209
Title: A PHASE I DOSE ESCALATION STUDY OF HYPOFRACTIONATED STEREOTACTIC RADIOTHERAPY WITH BEVACIZUMAB IN THE TREATMENT OF RECURRENT MALIGNANT GLIOMA
Brief Title: Hypofractionated Stereotactic Radiotherapy With Bevacizumab in the Treatment of Recurrent Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry); Columbia University (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-057
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Brain Cancer; MALIGNANT GLIOMA; Glioblastoma; Anaplastic Astrocytoma (AA); Anaplastic Oligodendroglioma (AO); Anaplastic Oligo-astrocytoma (AOA); Anaplastic Mixed Gliomas; Malignant Glioma NOS
Keywords: BEVACIZUMAB; HYPOFRACTIONATED STEREOTACTIC RADIOTHERAPY; Brain; CNS; anti-VEGF antibody; 11-057
MeSH Terms: conditions — Brain Neoplasms; Glioma; Glioblastoma; Astrocytoma; Oligodendroglioma | interventions — Bevacizumab; Radiosurgery

ARMS (1):
- Bevacizumab & Stereotactic Radiotherapy (Experimental): This will be a multicenter (MSKCC and UCSF) phase I dose escalation study to determine the maximum tolerated dose (MTD) of hypofractionated stereotactic radiotherapy when administered in combination with a fixed dose of bevacizumab.
  Interventions: Other: Bevacizumab & Stereotactic Radiotherapy

INTERVENTIONS:
Other: Bevacizumab & Stereotactic Radiotherapy — Treatment: (until treatment failure): bevacizumab 10 mg/kg IV once every two weeks on days 1 (+/- 3 days) and 15 (+/- 3 days) of every cycle (Cycle defined as 28 days). On day 28 (or up to 2 days before) of cycles 1 and 2 (and for every other cycle thereafter) patients will undergo a physical and radiological re-evaluation (MRI). Patients will begin stereotactic radiotherapy beginning anywhere from day 7 to day 10 of cycle 2 with escalating fraction sizes (interpatient - there is no intrapatient escalation). Assessment of response will be performed following cycles 1 and 2 then following every two cycles.

SUMMARY:
The best dose of radiation to be given with bevacizumab is currently unknown. This study will use higher doses of radiation with bevacizumab than have been used before. This study will test the safety of radiation given at different doses with bevacizumab to find out what effects, good and/or bad, it has on the patient and the malignant glioma or related brain cancers.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have EITHER
* Histologically confirmed intracranial malignant glioma of the following types: Glioblastoma, Anaplastic astrocytoma (AA), Anaplastic oligodendroglioma (AO), Anaplastic oligo-astrocytoma (AOA) also called anaplastic mixed gliomas, Malignant glioma NOS (not otherwise specified). Patients will be eligible if the original histology was low-grade glioma and a subsequent histological diagnosis of a high grade (malignant) glioma is made.

OR

* Histologically confirmed low grade (WHO grade II) gliomas (such as low grade astrocytoma, low grade oligodendroglioma, low grade oligo-astrocytoma (mixed gliomas), or low grade glioma NOS) IF there is radiographic evidence by MRI of malignant transformation but histologic confirmation of high grade (malignant) transformation would not be otherwise undertaken for routine clinical care. Inclusion of patients in this group will allow increased accrual rapidity by enrolling patients who are otherwise ineligible for almost all malignant glioma trials yet whom are treated presumptively for malignant glioma. The primary aim of the phase I study is not determination of efficacy. Therefore, inclusion of such patients will not affect efficacy analyses.

Participating site confirmation is adequate.

* Able to undergo brain MRI scans.
* MRI scan with gadolinium contrast showing geographically-circumscribed tumor ≤40 cc incorporating both enhancing and non-enhancing volume. This is calculated by the product of maximum measurements in 3 dimensions divided by 2. Tumors exceeding this limit may be eligible and any question should be directed to a Radiation Oncology Investigator and the MSK PI. (The MRI must be performed on a steroid dosage that has been stable or decreasing for at least 5 days. Patients on no steroids are eligible. If the steroid dose is increased between date of imaging and registration, a new baseline MRI is required).
* Prior treatment with approximately 60 Gy of radiotherapy.
* Patients must have recovered from the toxic effects of prior therapy including but not limited to:
* An interval of ≥ 4 weeks (28 days) from prior cytotoxic therapy except 6 weeks from nitrosoureas
* An interval of ≥ 1 week (7 days) from any non-cytotoxic agents
* An interval of ≥ 3 months from the completion of radiation therapy
* Absolute neutrophil count ≥ 1,500/mm3.
* Platelet count ≥ 100,000/mm3.
* Hemoglobin ≥ 10 g/dl.
* Serum creatinine ≤ 2 times upper limit of normal.
* Total bilirubin ≤ 2 times upper limit of normal.
* SGOT and SGPT both ≤ 3 times upper limit of normal.
* ≥18 years of age.
* Karnofsky Performance Score ≥ 60
* Life expectancy ≥ 12 weeks
* Men and women with reproductive potential must agree to use an acceptable method of birth control during treatment and for six months after completion of treatment.
* Written informed consent prior to registration on study.

Exclusion Criteria:

* Prior treatment with radiosurgery
* Prior disease progression/recurrence during or immediately following treatment with bevacizumab. Any question should be directed to the PI.
* Multicentric glioma
* Other malignancy (with the exception of cervical carcinoma in situ or basal cell carcinoma of the skin) for which there has been treatment within the last 3 years
* Serious medical or psychiatric illness that would in the opinion of the investigator interferes with the prescribed treatment.
* Pregnant or breast feeding women
* Inadequately controlled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure > 100 mmHg)
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* Grade 2 or greater congestive heart failure
* History of myocardial infarction, unstable angina, stroke, or transient ischemic attack within 12 months prior to Day 1
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
* History of hemoptysis ≥1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 of treatment or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Proteinuria as demonstrated by a UPC ratio ≥ 1.0 at screening
* Known hypersensitivity to any component of bevacizumab
* History of peptic ulcer within the last 6 months
* Clinically significant peripheral vascular disease
* Craniotomy wound that has not sufficiently healed
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Glioma showing prior spontaneous hemorrhage as determined from the clinical history or from any preoperative CT or MRI scan (excluding grade 1 punctate, incidentally found).
* Longest uni-dimensional measurement of contrast enhancing tumor ≥ 4cm. Tumors exceeding this limit may be eligible and any question should be directed to a Radiation Oncology Investigator and the MSK PI.
* Tumor must not invade the corpus callosum
* Tumor must not invade the brainstem
* Suspected or documented radionecrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-07-08 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
To establish the maximum tolerated dose (MTD) | 1 year
  of hypofractionated stereotactic re-irradiation delivered with concomitant bevacizumab in recurrent malignant gliomas (using a standard 3+3 design).

SECONDARY OUTCOMES:
Response rate | 1 year
  Median overall survival and progression-free survival, along with the estimated survival and PFS rates at specified time points will be estimated using Kaplan-Meier method. Confidence intervals will be included with all point estimates. Response rate will be estimated using an exact binomial distribution together with 95% confidence interval.
Median progression free survival | 1 year
  Median overall survival and progression-free survival, along with the estimated survival and PFS rates at specified time points will be estimated using Kaplan-Meier method. Confidence intervals will be included with all point estimates. Response rate will be estimated using an exact binomial distribution together with 95% confidence interval.
6 month progression-free survival rate | 1 year
  Median overall survival and progression-free survival, along with the estimated survival and PFS rates at specified time points will be estimated using Kaplan-Meier method. Confidence intervals will be included with all point estimates. Response rate will be estimated using an exact binomial distribution together with 95% confidence interval.
Median overall survival | 1 year
  Median overall survival and progression-free survival, along with the estimated survival and PFS rates at specified time points will be estimated using Kaplan-Meier method. Confidence intervals will be included with all point estimates. Response rate will be estimated using an exact binomial distribution together with 95% confidence interval.
Use of tractography to predict routes of progression in gliomas (MSKCC only) | 1 year
  DTI will be acquired at the time of the patient's routinely scheduled brain MRIs but at least on the baseline scan and the MRI 1 month after cycle 2. DTI parameters: A spin-echo echo-planar sequence using 25 gradient directions, TR/TE 11000/100 msec; matrix 128 × 128; in-plane resolution 1.88 × 1.88 mm; slice thickness 3 mm; b-value 1000 sec/mm2; NEX 1 and maximum diffusion gradient strength 22mTm-1.
Correlation of VEGF and VEGFR IHC and related pathways (MSKCC only) and MGMT promoter methylation with efficacy | 1 year
  Exploratory analyses related to VEGFR signaling including IHC for VEGF and VEGFR on pre-treatment tissue and post-treatment tissue and the analysis of biological correlate data has the overall goal of providing increased understanding of the nature of the response to bevacizumab but the amount of data available for the various measures is uncertain. Information may also be limited by the impact of intervening treatment between the most recent surgery and initiation of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kaley, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - University of California San Francisco, San Francisco, California
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Clarke J, Neil E, Terziev R, Gutin P, Barani I, Kaley T, Lassman AB, Chan TA, Yamada J, DeAngelis L, Ballangrud A, Young R, Panageas KS, Beal K, Omuro A. Multicenter, Phase 1, Dose Escalation Study of Hypofractionated Stereotactic Radiation Therapy With Bevacizumab for Recurrent Glioblastoma and Anaplastic Astrocytoma. Int J Radiat Oncol Biol Phys. 2017 Nov 15;99(4):797-804. doi: 10.1016/j.ijrobp.2017.06.2466. Epub 2017 Jun 30. PMID 28870792
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm